CLINICAL TRIAL: NCT00412750
Title: A Randomized, Open-label, Controlled, Multi-center Two-year Study Comparing Efficacy and Safety of Telbivudine, 600 mg PO in Combination With Peginterferon Alpha-2a sq 180 µg With Peginterferon Alpha-2a Monotherapy, and With Telbivudine Monotherapy in Treatment naïve Patients With HBeAg-positive CHB.
Brief Title: Efficacy and Safety of Telbivudine in Treatment naïve Patients With Hepatitis B e Antigen (HBeAg)-Positive Chronic Hepatitis B (CHB)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Enrollment stopped for safety issues
Sponsor: Novartis (Industry)
Responsible Party: novartis, novatis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600A2406; NCT00376389 (obsolete NCT alias)
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Results first posted 2011-07-13 (Estimated); Last update posted 2011-07-13 (Estimated); Status verified 2011-06

CONDITIONS: Hepatitis B
Keywords: hepatitis B; hepatitis B Virus (HBV); chronic hepatitis B; telbivudine; peginterferon
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic | interventions — Telbivudine; peginterferon alfa-2a

ARMS (3):
- LdT+ PEG-INF (Experimental): Telbivudine (LdT) 600 mg orally once a day for 104 weeks in combination with peginterferon alpha-2a (PEG-INF)180 μg subcutaneous injection once a week for 52 weeks.
  Interventions: Drug: Telbivudine (LdT); Drug: peginterferon alpha-2a
- LdT Monotherapy (Experimental): Telbivudine (LdT) monotherapy: 600 mg orally once daily for 104 weeks.
  Interventions: Drug: Telbivudine (LdT)
- PEG-INF Monotherapy (Active Comparator): Peginterferon alpha-2a (PEG- INF) monotherapy: 180 μg subcutaneous injection once a week for 52 weeks.
  Interventions: Drug: peginterferon alpha-2a

INTERVENTIONS:
Drug: Telbivudine (LdT) — 600 mg orally once daily for 104 weeks.
  Other Names: Sebivo
  Arms: LdT Monotherapy; LdT+ PEG-INF
Drug: peginterferon alpha-2a — 180 μg subcutaneous injection once a week for 52 weeks.
  Other Names: Pegasys
  Arms: LdT+ PEG-INF; PEG-INF Monotherapy

SUMMARY:
To evaluate the combination of telbivudine 600 mg orally (PO) once daily and peginterferon alpha-2a 180 ug subcutaneous (sq) injection weekly for antiviral efficacy in comparison to peginterferon alpha-2a monotherapy.

ELIGIBILITY:
Inclusion Criteria:

Documented Chronic hepatitis B (CHB) defined by all of the following:

* Clinical history compatible with CHB
* Detectable serum Hepatitis B Surface Antigen (HBsAg) at the Screening visit and at least 6 months prior
* HBeAg-positive at the Screening visit
* Hepatitis B 'e' Antibody (HBeAb)-negative at the Screening visit
* History of evidence of chronic liver inflammation,
* Elevated serum Alanine aminotransferase (ALT) level (1.3 - 10 x upper limit of normal (ULN)) at the Screening visit
* Serum HBV DNA level ≥ 6 log10 copies/mL,
* Chronic liver inflammation on previous liver biopsy within the previous 24 months.

Exclusion Criteria:

* Co-infection with Hepatitis C Virus (HCV), Hepatitis D Virus (HDV), or Human Immunodeficiency Virus (HIV).
* Has any of the following drug therapy:

  * Previously been treated in a trial with telbivudine
  * Received nucleoside or nucleotide therapy whether approved or investigational
  * Received any immunomodulatory treatment in the 12 months before Screening for this study.
  * Has a medical condition that required prolonged or frequent use of systemic acyclovir or famciclovir.
  * Has a medical condition that requires frequent or prolonged use of systemic corticosteroids although inhaled or intra-articular corticosteroids are allowed.
  * Has a medical condition requiring the chronic or prolonged use of potentially hepatotoxic drugs or nephrotoxic drugs.
  * Is currently abusing alcohol or illicit drugs or has a history of alcohol abuse illicit substance abuse within the preceding two years.
  * Uses other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
  * Is currently receiving methadone.
* Patient has any of the following:

  * History of or clinical signs/symptoms of hepatic decompensation such as ascites, esophageal variceal bleeding, hepatic encephalopathy, or spontaneous bacterial peritonitis.
  * History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin. Patients with previous findings suggestive of possible HCC should have the disease ruled out prior to entrance into the study.
  * One or more additional known primary or secondary causes of liver disease other than hepatitis B, including steatohepatitis.
  * History of clinical and laboratory evidence of chronic pancreatitis, or demonstrates a clinical and laboratory course consistent with current pancreatitis.
* Has laboratory values during screening visit not within normal limits.
* Is pregnant or breastfeeding.
* Is a women of child-bearing potential that is unwilling to practice birth control.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2006-12; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Novartis, San Francisco, California, United States

REFERENCES:
- [Derived] Marcellin P, Wursthorn K, Wedemeyer H, Chuang WL, Lau G, Avila C, Peng CY, Gane E, Lim SG, Fainboim H, Foster GR, Safadi R, Rizzetto M, Manns M, Bao W, Trylesinski A, Naoumov N. Telbivudine plus pegylated interferon alfa-2a in a randomized study in chronic hepatitis B is associated with an unexpected high rate of peripheral neuropathy. J Hepatol. 2015 Jan;62(1):41-7. doi: 10.1016/j.jhep.2014.08.021. Epub 2014 Aug 23. PMID 25152207

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a randomized, open-label, controlled, multi-center two-year study enrolling male and female subjects starting December 2006 and ending February 2009.
Groups:
- LdT + PEG-INF: Telbivudine (LdT) 600 mg orally once a day for 104 weeks in combination with peg interferon (PEG-INF) alpha-2a 180 μg subcutaneous injection once a week for 52 weeks.
- PEG-INF Monotherapy: Peg interferon (PEG- INF) alpha-2a monotherapy: 180 μg subcutaneous injection once a week for 52 weeks.
Period: Overall Study
Arm/Group | LdT + PEG-INF | LdT Monotherapy | PEG-INF Monotherapy
Started | 50 | 55 | 54
Completed | 19 | 34 | 31
Not Completed | 31 | 21 | 23
Not completed — Abnormal laboratory value(s) | 1 | 0 | 0
Not completed — Administrative problems | 21 | 17 | 14
Not completed — Adverse Event | 8 | 3 | 3
Not completed — Lost to Follow-up | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LdT + PEG-INF | LdT Monotherapy | PEG-INF Monotherapy | Total
Number analyzed (Participants) | 50 | 55 | 54 | 159
Age Continuous [Mean (Standard Deviation); unit: years] | 35.6 (10.00) | 35.0 (11.48) | 33.8 (9.47) | 34.7 (10.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 15 | 20 | 51
  Male | 34 | 40 | 34 | 108

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved HBV DNA Non-detectability With Peginterferon Alpha-2a Plus Telbivudine Combination Therapy Versus Peginterferon Alpha-2a Monotherapy
Description: The original primary efficacy variable was the percentage of patients achieving HBV DNA non-detectability utilizing polymerase chain reaction (PCR) (threshold for detection 300 copies/mL); however, this analysis was not performed due to premature study termination.
Time Frame: At week 52
Population: The analysis was planned on intention to treat (ITT) population. Due to premature study termination, the analysis was not performed.
Measure: Number; unit: Percentage of participants
Arm/Group | LdT + PEG-INF | PEG-INF Monotherapy
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline in HBV DNA Concentration
Description: The change from baseline in HBV DNA concentration at Weeks 12 and 24 was analyzed using an analysis of covariance (ANCOVA) model with baseline HBV DNA concentration (log10 copies/ml) as a covariate, treatment and country as factors.
Time Frame: Weeks 12 and 24
Population: Intent to Treat (ITT) population. n= the number of patients who have both baseline and post baseline observation for the respective week
Measure: Least Squares Mean (Standard Error); unit: log 10 copies/ml
Arm/Group | LdT + PEG-INF | LdT Monotherapy | PEG-INF Monotherapy
Number analyzed (Participants) | 49 | 53 | 53
log 10 copies/ml
  Week 12 (n= 37, 52, 50) | -6.0569 (0.3124) | -5.1658 (0.2717) | -1.8991 (0.2607)
  Week 24 (n= 17, 48, 42) | -6.9187 (0.5462) | -5.9633 (0.3523) | -2.4513 (0.3485)

3. Secondary Outcome: Percentage of Participants Who Experienced Virologic Breakthrough at Weeks 48 and 52
Description: The percentage of participants with Virologic breakthrough at Week 48 and 52 by treatment. For the subgroup of patients on treatment who achieve HBV DNA >= 1 log10 copies/mL reduction from baseline on 2 consecutive visits, Virologic Breakthrough is defined as HBV DNA >= 1 log10 copies/mL from nadir on two consecutive visits.
Time Frame: Weeks 48 and 52
Population: Intent to treat (ITT) population. As most patients did not reach Week 48 and Week 52, the LOCF was used.
Measure: Number; unit: Percentage of participants
Arm/Group | LdT + PEG-INF | LdT Monotherapy | PEG-INF Monotherapy
Number analyzed (Participants) | 49 | 53 | 53
Percentage of participants
  Virologic breakthrough Week 48 | 0.0 | 5.7 | 7.5
  Virologic breakthrough Week 52 | 0.0 | 7.5 | 9.4

4. Secondary Outcome: Percentage of Participants With Hepatitis B 'e' Antigen (HBeAg) Loss and HBeAg Seroconversion
Description: HBeAg loss is defined as the loss of detectable serum HBeAg in a patient who was HBeAg positive at baseline. HBeAg seroconversion is defined as HBeAg loss with detectable Hepatitis B 'e' antibody (HBeAb). The efficacy was assessed for 18 weeks, 24 weeks, 48 weeks, 52 weeks and on treatment completion (TC).
Time Frame: Weeks 18, 24, 48, 52 and Treatment completion (TC)
Population: Intent to Treat (ITT) population. The study was terminated and some participants did not complete all visits. "n" in each of the categories represents the number of participants in each arm with non-missing efficacy endpoint observations for the respective week and on treatment completion (TC).
Measure: Number; unit: Percentage of participants
Arm/Group | LdT + PEG-INF | LdT Monotherapy | PEG-INF Monotherapy
Number analyzed (Participants) | 49 | 53 | 53
Percentage of participants
  HBeAg loss Week 18 (n=28,51,45) | 17.9 | 7.8 | 8.9
  HBeAg seroconversion Week 18 (n=28,51,45) | 17.9 | 7.8 | 8.9
  HBeAg loss Week 24 (n=17,48,42) | 17.6 | 6.3 | 11.9
  HBeAg seroconversion Week 24 (n=17,48,42) | 7.6 | 4.2 | 11.9
  HBeAg loss Week 48 (n=0,19,12) | NA — Participants in the LdT + PEG-INF arm were discontinued prior to week 48, hence no data is available | 36.8 | 25.0
  HBeAg seroconversion Week 48 (n=0,19,12) | NA — Participants in the LdT + PEG-INF arm were discontinued prior to week 48, hence no data is available | 36.8 | 25.0
  HBeAg loss Week 52 (n=0,10,6) | NA — Participants in the LdT + PEG-INF arm were discontinued prior to week 48, hence no data is available | 50.0 | 16.7
  HBeAg seroconversion Week 52 (n=0,10,6) | NA — Participants in the LdT + PEG-INF arm were discontinued prior to week 48, hence no data is available | 50.0 | 16.7
  HBeAg loss TC (n=14,24,9) | 7.1 | 29.2 | 33.3
  HBeAg seroconversion TC (n=14,24,9) | 7.1 | 25.0 | 33.3

5. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA Non-detectability With Telbivudine Monotherapy Versus Peginterferon Alpha-2a Monotherapy
Description: Antiviral efficacy was assessed by percentage of patients achieving HBV DNA non-detectability assay utilizing polymerase chain reaction (PCR) (threshold for detection 300 copies/mL); however, this analysis was not performed due to premature study termination.
Time Frame: Week 52
Population: The analysis was planned on intent to treat (ITT) population. Due to premature study termination, the analysis was not performed.
Measure: Number; unit: Percentage of participants
Arm/Group | LdT Monotherapy | PEG-INF Monotherapy
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA Non-detectability With Peginterferon Alpha-2a Plus Telbivudine Combination Therapy Versus Telbivudine Monotherapy
Description: as for outcome 5
Time Frame: Week 52
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | LdT + PEG-INF | LdT Monotherapy
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Percentage of Participants With HBV DNA Non-detectability and Alanine Aminotransferase (ALT) Normalization at Week 12 and Week 24 in Participants With HBeAg-positive Chronic Hepatitis B (CHB)
Description: The percentage of participants who achieved HBV DNA non-detectability using the COBAS Amplicor HBV Monitor assay utilizing polymerase chain reaction (PCR) (threshold for detection 300 copies/mL) and Alanine aminotransferase (ALT) normalization defined as ALT within normal limits on two successive visits for a patient with an elevated ALT (>1.0 x upper limit normal) at baseline summarized at Weeks 12 and 24.
Time Frame: Weeks 12 and 24
Population: Intent to Treat (ITT) population. The study was terminated and some participants did not complete all visits. "n" in each of the categories represents the number of participants in each arm with non-missing efficacy endpoint observations for the respective week.
Measure: Number; unit: Percentage of participants
Arm/Group | LdT + PEG-INF | LdT Monotherapy | PEG-INF Monotherapy
Number analyzed (Participants) | 49 | 53 | 53
Percentage of participants
  HBV DNA non-detectability Week 12 (n=37,52,50) | 13.5 | 9.6 | 0.0
  ALT normalization Week 12 (n=37,52,50) | 13.5 | 28.8 | 20.0
  HBV DNA non-detectability Week 24 (n=17,48,42) | 70.6 | 35.4 | 7.1
  ALT normalization Week 24 (n=17,48,41) | 11.8 | 54.2 | 31.7

ADVERSE EVENTS:
Description: Safety Population defined as all patients who received one dose of study drug and had at least one post baseline assessment.
Arm/Group | LdT + PEG-INF | LdT Monotherapy | PEG-INF Monotherapy
Serious Adverse Events (participants affected / at risk) | 11/50 | 2/54 | 2/54
Other Adverse Events (participants affected / at risk) | 38/50 | 35/54 | 47/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LdT + PEG-INF (N=50) | LdT Monotherapy (N=54) | PEG-INF Monotherapy (N=54)
Mitochondrial myopathy (Congenital, familial and genetic disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 3 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0
Depression suicidal (Psychiatric disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LdT + PEG-INF (N=50) | LdT Monotherapy (N=54) | PEG-INF Monotherapy (N=54)
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 5
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 4
Tinnitus (Ear and labyrinth disorders) | 1 | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 6 | 3 | 4
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 3
Nausea (Gastrointestinal disorders) | 10 | 4 | 9
Vomiting (Gastrointestinal disorders) | 2 | 1 | 3
Asthenia (General disorders) | 8 | 6 | 10
Fatigue (General disorders) | 8 | 3 | 7
Influenza like illness (General disorders) | 8 | 2 | 12
Irritability (General disorders) | 2 | 2 | 4
Pain (General disorders) | 3 | 2 | 4
Pyrexia (General disorders) | 11 | 2 | 13
Influenza (Infections and infestations) | 1 | 2 | 5
Nasopharyngitis (Infections and infestations) | 0 | 4 | 2
Sinusitis (Infections and infestations) | 0 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 4 | 11 | 10
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 3
Weight decreased (Investigations) | 3 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 5 | 3 | 4
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 5 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4
Headache (Nervous system disorders) | 8 | 9 | 17
Lethargy (Nervous system disorders) | 3 | 0 | 2
Paraesthesia (Nervous system disorders) | 6 | 0 | 2
Anxiety (Psychiatric disorders) | 3 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 5
Insomnia (Psychiatric disorders) | 3 | 2 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 3 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 2 | 15
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 9
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.